CLINICAL TRIAL: NCT00569075
Title: Apoptotic Biomarkers of Periodontal Disease
Brief Title: Apoptic Biomarkers of Periodontal Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Yvonne Kapila, University of Michigan
Other Study IDs: 2004-04
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Periodontitis
Keywords: Apoptic biomarkers; Early detection periodontitis; Gingival crevicular fluid; Healthy subjects
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva and plaque
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High Risk: High risk disease prone population
  Interventions: Other: collection of gingival crevicular fluid
- Low Risk: Low risk disease population
  Interventions: Other: collection of gingival crevicular fluid

INTERVENTIONS:
Other: collection of gingival crevicular fluid — GCF samples will be collected at 3 month intervals

SUMMARY:
The goal of this study is to facilitate early diagnosis of gum disease. Proteins associated with cell death will be isolated from gum pockets of diseased and healthy patients and evaluated.

DETAILED DESCRIPTION:
Early detection of the progression of periodontitis is difficult because it typically relies on comparisons of clinical measurements made with a calibrated probe and nonstandardized radiographs over time. Both methods detect periodontal breakdown only after it has occurred. Therefore, considerable emphasis has been placed on identifying more specific and sensitive methods to diagnose and detect periodontal disease progression. The overall goal of this project is to determine whether specific apoptosis-associated proteins, specifically fibronectin (FN) fragments, caspase-3, soluble Fas, and soluble Fas ligand, sampled from gingival crevicular fluid (GCF) can be used as markers for periodontal disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age of 18
* Healthy or diagnosis of periodontitis

Exclusion Criteria:

* Active treatment with anti-inflammatory agents such as NSAIDs or steroids and pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults with healthy gums or those with periodontitis
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Kapila, DDS, PhD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States